CLINICAL TRIAL: NCT04692103
Title: Serial [F-18] Fluoroestradiol (FES) PET Imaging to Evaluate Endocrine-targeted Therapy
Brief Title: Serial FES PET/CT to Measure Hormone Expression in Patients Undergoing Endocrine Targeted Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Delphine Chen, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RG1007834; 10465 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Estrogen Receptor Positive; Primary or Recurrent Breast Carcinoma; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — 16-fluoroestradiol; Magnetic Resonance Spectroscopy; X-Rays; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (F-18 FES PET/CT) (Experimental): Patients undergo F-18 FES PET/CT scan at baseline. Patients also undergo F-18 FES PET/CT and FDG PET/CT between 1-12 weeks after starting therapy, and then 1-12 weeks after the second FES PET/CT scan. Repeat FDG PET may be omitted in patients on selective estrogen receptor degrader.
  Interventions: Drug: F-18 16 Alpha-Fluoroestradiol; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Drug: Fludeoxyglucose F-18; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: F-18 16 Alpha-Fluoroestradiol — Undergo F-18 FES PET/CT
  Other Names: F-18 FES; FES; Fluorine-18 16 alpha-fluoroestradiol; Fluoroestradiol F-18
Procedure: Positron Emission Tomography — Undergo F-18 FES PET/CT
  Other Names: Medical Imaging; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography
Procedure: Computed Tomography — Undergo F-18 FES PET/CT
  Other Names: CAT Scan; Computerized Axial Tomography; CT scan
Drug: Fludeoxyglucose F-18 — Undergo FDG PET/CT
  Other Names: FDG; Fluorodeoxyglucose F18; 18FDG
Procedure: Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: Medical Imaging; PET; PET Scan
Procedure: Computed Tomography — Undergo FDG PET/CT
  Other Names: CAT Scan
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial studies use of F-18 16 alpha-fluoroestradiol ([F-18] FES) positron emission tomography (PET)/computed tomography (CT) in measuring tumor hormone receptor expression in patients undergoing endocrine-targeted therapy for newly diagnosed breast cancer or breast cancer that has come back or spread to other places in the body. Comparing results of diagnostic procedures done before, during, and after hormone therapy may help measure a patient's response to treatment.

DETAILED DESCRIPTION:
OUTLINE:

Patients undergo F-18 FES PET/CT scan at baseline. Patients also undergo F-18 FES PET/CT and FDG PET/CT between 1-12 weeks after starting therapy, and then 1-12 weeks after the second FES PET/CT scan. Repeat FDG PET may be omitted in patients on selective estrogen receptor degrader.

After completion of study, patients are followed up for up to 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult, non-pregnant patients with biopsy-proven or clinically obvious primary, recurrent or metastatic breast cancer
* Breast cancer from ER+ primary that is seen on other imaging tests. Tumor ER expression must have been confirmed by immunohistocytochemistry of primary tumor or recurrent disease.
* At least one site of disease 1.5 cm or greater is needed to meet the spatial resolution limits of PET imaging.
* Patients must have been off tamoxifen or other estrogen receptor blocking agents for at least 6 weeks and off chemotherapy for 3 weeks for the initial baseline FES.
* Patients must be selected for an endocrine targeted therapy regimen for treatment of their breast cancer by the referring oncologist. Selected treatments may be part of experimental treatment protocols for which the patient would be separately consented.
* Patients must be willing to undergo serial imaging procedures.
* Patients must agree to allow access to clinical records regarding response to treatment and long term follow up.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* An inability to lie still for the tests
* Individuals weighing more than 300 lb. (this is the weight limit of the scanner table)
* Pregnant or lactating. Women of childbearing potential with either a positive or no pregnancy test at baseline are excluded.
* Any other life-threatening illness (e.g. serious, uncontrolled concurrent infection or clinically significant cardiac disease - congestive heart failure, symptomatic coronary artery disease, cardiac arrhythmia not well controlled with medication).
* Use of tamoxifen, faslodex, DES or any other ER blocking agent < 6 weeks or chemotherapy < 3 weeks prior to imaging scan.
* Uncontrolled diabetes mellitus (fasting glucose > 200 mg/dL)
* Adult patients who require monitored anesthesia for PET scanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2041-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (F-18 FES PET/CT): Patients undergo F-18 FES PET/CT scan at baseline. Patients also undergo F-18 FES PET/CT and FDG PET/CT between 1-12 weeks after starting therapy. Repeat FDG PET may be omitted in patients on selective estrogen receptor degrader.
Period: Overall Study
Arm/Group | Diagnostic (F-18 FES PET/CT)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (F-18 FES PET/CT)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 71 [70 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in F-18 16 Alpha-fluoroestradiol (FES) Standardized Uptake Value (SUV) - Avg SULmax
Description: FES uptake will be quantified using lean body mass adjusted SUV (SUL). Percentage change in FES average SULmax between baseline and a second FES scan will be calculated for up to 3 lesions per patient.
Time Frame: From time of first F-18 FES-PET/CT scan to time of second F-18 FES-PET/CT scan (approximately 1-12 weeks)
Population: 2 patients had 2 FES scans each
Measure: Mean (Full Range); unit: Percentage decrease in avgSUL
Arm/Group | Diagnostic (F-18 FES PET/CT)
Number analyzed (Participants) | 2
Percentage decrease in avgSUL | 78 [77 to 79]

2. Primary Outcome: F-18 16 Alpha-fluoroestradiol (FES) Uptake
Description: Quantitative measures of FES uptake for each disease site will be determined by drawing regions-of-interest on lesions to determine maximal FES uptake (SUVmax) per lesion. Up to 10 sites seen on the static torso survey will be quantified.
Time Frame: From time of first F-18 FES-PET/CT scan to time of second F-18 FES-PET/CT scan (approximately 1-12 weeks)
Population: 2 patients had 2 scans each
Measure: Mean (Full Range); unit: average SUVmax
Arm/Group | Diagnostic (F-18 FES PET/CT)
Number analyzed (Participants) | 2
average SUVmax
  FES scan 1 | 5.7 [4.6 to 6.8]
  FES scan 2 | 1.4 [1.0 to 1.7]

3. Primary Outcome: Proportion of Patients With a Threshold of Percentage Change, or That Surpass a Targeted Follow-up F-18 16 Alpha-fluoroestradiol (FES) Standardized Uptake Value (SUV)
Description: The number of patients showing a 20% increase in FES uptake (SULmean or SUVmax) compared to baseline from the first to second scan using a 90% Wilson score binomial confidence interval.
Time Frame: From time of first F-18 FES-PET/CT scan to time of second F-18 FES-PET/CT scan (approximately 1-12 weeks)
Population: 2 patients had 2 FES scans each
Measure: Number; unit: participants with increased FES uptake
Arm/Group | Diagnostic (F-18 FES PET/CT)
Number analyzed (Participants) | 2
participants with increased FES uptake | 0

4. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression will be measured as the time from the start of endocrine therapy to the time the patient is first recorded as having disease progression.
Time Frame: From start of therapy up to 20 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 hours after each FES PET/CT study (the time-frame of F18-FES decay)
Arm/Group | Diagnostic (F-18 FES PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT04692103/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT04692103/ICF_001.pdf